CLINICAL TRIAL: NCT05009862
Title: The Impact of Factor Xa Inhibition on Thrombosis, Platelet Activation, and Endothelial Function in Peripheral Artery Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Aaron W. Aday, MD, MSc, Assistant Professor Division of Cardiovascular Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200447; 5K23HL151871 (NIH)
Record Dates: First submitted 2021-07-09; First posted 2021-08-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Artery Disease; PAD; Thrombosis; Rivaroxaban; Anticoagulant
MeSH Terms: conditions — Peripheral Arterial Disease; Thrombosis | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Participants will receive 81mg daily of aspirin + placebo for 30 days.
  Interventions: Drug: Placebo; Drug: Aspirin 81Mg Ec Tab
- Intervention (Experimental): Participants will receive 81mg of aspirin + rivaroxaban 2.5mg twice daily for 30 days.
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet; Drug: Aspirin 81Mg Ec Tab

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — rivaroxaban 2.5 milligrams twice daily
  Arms: Intervention
Drug: Placebo — placebo
  Arms: Control
Drug: Aspirin 81Mg Ec Tab — aspirin 81 milligrams

SUMMARY:
The purpose of this study is to understand how the drug rivaroxaban improves symptoms associated with peripheral artery disease.

DETAILED DESCRIPTION:
The Primary Investigator's central hypothesis is that activation of thrombotic pathways and downstream effectors of factor Xa signaling contribute to the development of PAD and its complications.

Aim 1: To assess the impact of rivaroxaban on macrovascular endothelial function in a randomized, double-blind, placebo-controlled crossover intervention in humans with PAD.

Aim 2: To assess the impact of rivaroxaban on PAR-1-mediated platelet activation in addition to its pleiotropic effects on thrombosis, thrombolysis, and inflammation in a randomized, double-blind, placebo-controlled crossover intervention in humans with PAD.

ELIGIBILITY:
Inclusion criteria:

History of peripheral artery disease (PAD) defined as:

* Previous aorto-femoral bypass surgery, limb bypass surgery, or percutaneous transluminal angioplasty revascularization of the iliac or infra-inguinal arteries, or
* Previous limb or foot amputation for arterial vascular disease, or
* An ankle/arm blood pressure (BP) ratio less than 0.90, or
* Significant peripheral artery stenosis (≥50%) documented by angiography, or by duplex ultrasound, or
* An ankle-brachial index (ABI) greater than 1.4 with a toe-brachial index (TBI) less than 0.7 AND
* Willing and able to provide written informed consent
* Receiving aspirin therapy prior to enrollment

Exclusion Criteria:

* High risk of bleeding
* Stroke within 1 month of any history of hemorrhagic or lacunar stroke
* Severe heart failure with known ejection fraction less than 30% or New York Heart Association (NYHA) class III or IV symptoms
* Estimated glomerular filtration rate less than 15 mL/min/1.73m2
* Need for dual-antiplatelet therapy, other non-aspirin antiplatelet therapy, or oral anticoagulant therapy
* Known non-cardiovascular disease that is associated with poor prognosis (e.g. metastatic cancer) or that increases the risk of an adverse reaction to study interventions
* History of hypersensitivity or known contraindication to rivaroxaban or aspirin
* Systemic treatment with strong inhibitors of both CYP 3A4 and p-glycoprotein (e.g. systemic azole antimycotics, such as ketoconazole, and human immunodeficiency virus [HIV]-protease inhibitors, such as ritonavir), or strong inducers of CYP 3A4, i.e. rifampicin, rifabutin, phenobarbital, phenytoin, and carbamazepine
* Any known hepatic disease associated with coagulopathy
* Subjects who are pregnant, breastfeeding, or are of childbearing potential, and sexually active and not practicing an effective method of birth control (e.g. surgically sterile, prescription oral contraceptives, contraceptive injections, intrauterine device, double- barrier method, contraceptive patch, male partner sterilization)
* Concomitant participation in another study with investigational drug
* Upcoming invasive procedure within 3 months
* Invasive procedure within the prior 1 month
* Being treated for an active infection
* Acute or chronic limb-threatening ischemia
* Known contraindication to any study related procedures

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Endothelium-dependent, flow-mediated dilation (FMD) of the brachial artery | Baseline to 37 days
  FMD will be measured by forearm high-resolution ultrasonography after treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
Endogenous PAR-1 activation as measured by flow cytometry | Baseline to 37 days
  Endogenous PAR-1 activation, a novel marker of platelet activation, will be measured by flow cytometry, following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo. The unit of measure will be relative fluorescence.

SECONDARY OUTCOMES:
Prothrombin time | Baseline to 37 days
  Prothrombin time will be measured using turbidimetric assays following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo. The unit of measure will be in seconds.
Partial thromboplastin time | Baseline to 37 days
  Partial thromboplastin time will be measured using turbidimetric assays following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo. The unit of measure will be seconds.
von Willebrand factor (vWF) | Baseline to 37 days
  Blood levels of von Willebrand factor will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
D-Dimer | Baseline to 37 days
  Blood levels of D-dimer will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
High-sensitivity C-reactive protein. | Baseline to 37 days
  Blood levels of high-sensitivity C-reactive protein will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo. The unit of measure will be mg/L.
Tumor necrosis factor-alpha | Baseline to 37 days
  Blood levels of tumor necrosis factor-alpha will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
Interleukin-1beta | Baseline to 37 days
  Blood levels of interleukin-1beta will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
Interleukin-6 | Baseline to 37 days
  Blood levels of interleukin-6 will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
Soluble intercellular adhesion molecule-1 (slCAM-1) | Baseline to 37 days
  Blood levels of soluble intercellular adhesion molecule-1 (slCAM-1) will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
Monocyte chemoattractant protein-1 (MCP-1) | Baseline to 37 days
  Blood levels of monocyte chemoattractant protein-1 (MCP-1) will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
Plasminogen activator inhibitor 1 (PAI-1) | Baseline to 37 days
  Blood levels of plasminogen activator inhibitor 1 (PAI-1) will be measured following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
CD41a (Integrin alpha-II-beta) | Baseline to 37 days
  CD41a, a marker of platelet activation, will be measured by flow cytometry following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.
CD62p (P-Selectin) | Baseline to 37 days
  CD62p, a marker of platelet activation, will be measured by flow cytometry following treatment with low-dose rivaroxaban plus aspirin and compared to the baseline value following treatment with aspirin plus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron W Aday, MD, Principal Investigator — VUMC Cardiovascular Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No